CLINICAL TRIAL: NCT04062071
Title: Prevalence of Use of Anticoagulant, and Associated Factors of Anticoagulant Refusal in Non-valvular Atrial Fibrillation Patients---- A Study in Hong Kong General Out-patient Clinic
Brief Title: Use of Anticoagulant, and Associated Factors of Anticoagulant Refusal Atrial Fibrillation Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, chen liujing, resident, Prince of Wales Hospital, Shatin, Hong Kong
Other Study IDs: version1 last update 30/7/2019
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
Keywords: anticoagulants
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Atrial fibrillation is a clinically significant cardiac arrhythmia that increases the risk of stroke by 3 to 4 times. Oral anticoagulation has been shown to mitigate stroke risk by two-thirds among patients with AF and is widely recommended in optimizing AF management.Direct oral anticoagulants have also been demonstrated to be superior to warfarin with respect to the risk of fatal bleeding and stroke prevention.

However, the previous study finding highlighted a great gap between current guidelines and the clinical management of AF .Nonetheless, the decision for anticoagulant use is not straightforward.It is worth to investigate the updated prevalence of anticoagulant use, the reasons for not receiving anticoagulant, and the factors independently associated with anticoagulant refusal in patients with non-valvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis as atrial fibrillation
* aged ≧18 years
* able to given consent

Exclusion Criteria:

* Unable/unwillingness to sign informed consent to study
* mechanical heart valve
* moderate-to-severe mitral stenosis
* Transient atrial fibrillation from reversible cause (e.g., during respiratory tract infection or bronchospasm)
* pregnancy
* hospitalization within 1 month prior to inclusion in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all of the documented atrial fibrillation patients having regular follow up in GOPC in the study period
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-08-23 (Estimated); Primary Completion 2020-03-23 (Estimated); Study Completion 2020-03-23 (Estimated)

PRIMARY OUTCOMES:
The prevalence of anticoagulant use in non-valvular atrial fibrillation patients | August 2019 to March 2020
  calculate the prevalence of anticoagulant use in non-valvular atrial fibrillation patients

SECONDARY OUTCOMES:
the rate of the refusal of anticoagulant use | August 2019 to March 2020
  calculate the rate of refusal of anticoagulant use in the eligible non-valvular atrial fibrillation patients

CONTACTS AND LOCATIONS:
Locations (1):
- LIAO, Jiawei, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
no Conflict of interest